CLINICAL TRIAL: NCT01577381
Title: A Phase 2 Multi-center, Randomized, Double-masked, Placebo-controlled, Multi-dose Study To Investigate The Efficacy, Safety, Pharmacokinetics And Pharmacodynamics Of Rn6g (Pf-04382923) In Subjects With Geographic Atrophy Secondary To Age-related Macular Degeneration
Brief Title: Efficacy, Safety And Tolerability Study Of RN6G In Subjects With Geographic Atrophy Secondary to Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1181003; 2012-000823-42 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Age-Related Maculopathy
Keywords: Phase 2; Advanced Dry Age-Related Macular Degeneration; Geographic Atrophy; RN6G
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04382923 (Experimental)
  Interventions: Biological: RN6G
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RN6G — Intravenous, 11 doses, 30 minute infusion, dose ranging from 2.5 mg/kg up to a maximum of 15 mg/kg
  Arms: PF-04382923
Biological: Placebo — Intravenous, 11 doses, 30 minute infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of multiple doses of RN6G in subjects with Geographic Atrophy Secondary to Age-related Macular Degeneration.

DETAILED DESCRIPTION:
The trial was terminated early on April 12, 2013 due to an organizational decision, which was not based on safety or efficacy concerns. Subjects who were already enrolled into the study were followed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 60 and 90 years.
* Diagnosis of a geographic atrophy (GA) secondary to dry Age-Related Macular Degeneration.
* Best Corrected Visual Acuity (BCVA) of 20/80 or better in the study eye

Exclusion Criteria:

* Evidence of ocular disease other than geographic atrophy (GA) secondary to dry Age-Related Macular Degeneration in the study eye.
* History or diagnosis of exudative (wet) Age-Related Macular Degeneration, with subretinal or choroidal neovascular lesions in the study eye.
* Presence of disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, central nervous, immune, or gastrointestinal system

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (82):
  - Scottsdale Medical Imaging, Phoenix, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Premier Research Group Limited, Phoenix, Arizona
  - Radiology Limited, Tucson, Arizona
  - Retina Associates, Tucson, Arizona
  - Reeds Compounding Pharmacy, Tucson, Arizona
  - Methodist Hospital of Southern California, Arcadia, California
  - Retina Institute of California, Arcadia, California
  - Mink Radiologic Imaging, Beverly Hills, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Valley Radiology Medical Associates, Inc., Mountain View, California
  - Fairmount Pharmacy, Pasadena, California
  - Radiological Associates of Sacramento Medical Group, Inc. (MRI Imaging Only), Roseville, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Leiter's Compounding Pharmacy, San Jose, California
  - Cardiology Specialist of Orange County (ECG Evaluation Only), Santa Ana, California
  - Kenneth L. Nudleman M.D. (Neurology Exam Only), Santa Ana, California
  - Open Advantage MRI (Brain MRI Only), Santa Ana, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Quest Diagnostics Patient Service Center (Blood Draw Lab only), Santa Ana, California
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Maitland Avenue Urgent Care (Physical and Neurologic Exams Only), Altamonte Springs, Florida
  - Mid Florida Imaging (MRI Only), Altamonte Springs, Florida
  - Center for Retina and Macular Disease, Lakeland, Florida
  - Medeye Associates, Miami, Florida
  - Open MRI & CT of South Miami, Miami, Florida
  - Retina Care Specialists, LLP, Palm Beach Gardens, Florida
  - Premiere Research Institute At Palm Beach Neurology (MRI, Physical Exam, and Neurological Exam Only), West Palm Beach, Florida
  - Sabates Eye Center Research Division, Leawood, Kansas
  - O'Brien Pharmacy (Drug Shipment Only), Mission, Kansas
  - Diagnostic Imaging (MRI Only), Overland Park, Kansas
  - Apothecary By Design, Portland, Maine
  - Charles Cathcart M.D., Portland, Maine
  - Maine Eye Center, Portland, Maine
  - Intermed Diagnostic Imaging, South Portland, Maine
  - Advanced Open MRI, Toms River, New Jersey
  - Retina Vitreous Center, Toms River, New Jersey
  - Shore Neurology, PA, Toms River, New Jersey
  - King's Pharmacy, Brooklyn, New York
  - Zwager - Pesiri Radiology Group - MRI Exam Facility Only, East Setauket, New York
  - Advanced Neurological Care, PC - Neurology Exam Facility Only, Lynbrook, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Zwager - Pesiri Radiology Group - MRI Exam Facility Only, Merrick, New York
  - Lenox Hill Radiology/Regency Medical Imaging (MRI Only), New York, New York
  - Macula Care, Pllc, New York, New York
  - Lenox Hill Radiology (MRI Only), New York, New York
  - Zwager - Pesiri Radiology Group - MRI Exam Facility Only, Plainview, New York
  - Cardiology Consultants of Long Island, PC- Physical Exam Facility Only, Rockville Centre, New York
  - Advanced Neurological Care, PC - Neurology Exam Facility Only, Valley Stream, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Pro Scan Imaging, Mason, Ohio
  - Associates in Ophthalmology, Ltd., West Mifflin, Pennsylvania
  - UPMC West Mifflin (MRI Only), WestMifflin, Pennsylvania
  - Hawthorne Pharmacy, Columbia, South Carolina
  - InMed (MRI Facility), Columbia, South Carolina
  - Jay Markowitz, MD and Associates (Physical Exams Only), West Columbia, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - South Carolina Neurological Clinic (Neurological Exams Only), West Columbia, South Carolina
  - Centennial Medical Center (MRI Only), Nashville, Tennessee
  - Tennessee Retina, P.C, Nashville, Tennessee
  - Radiology Associates of North Texas, Arlington, Texas
  - Innovative Infusion, Arlington, Texas
  - Texas Retina Associates, Arlington, Texas
  - Kevin E. Conner, Arlington, Texas
  - Brian B. Berger, MD, PA, Austin, Texas
  - Retina Research Center, Austin, Texas
  - River Ranch Radiology, Austin, Texas
  - Sleep Medicine Consultants, Austin, Texas
  - Specialty Compounding, Cedar Park, Texas
  - Advanced Radiology Services, Edinburg, Texas
  - Edinburg Family Pharmacy, Edinburg, Texas
  - McAllen Advanced Medical Imaging, McAllen, Texas
  - McAllen Surgical Specialty Center, McAllen, Texas
  - Tommy Yee MD, McAllen, Texas
  - Valley Retina Institute,P.A., McAllen, Texas
  - Weslaco Advanced Imaging, Weslaco, Texas
  - Proliance Surgeons, Inc. PS DBA Vitreo Retinal Associates, Bellevue, Washington
  - Sound Prescriptions LLC, Bellevue, Washington
  - Orthopedic Physician Assoc. - MRI, Seattle, Washington
  - Proliance Surgeons, Inc. PS DBA Vitreo Retinal Associates, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1181003&StudyName=Efficacy%2C%20Safety%20And%20Tolerability%20Study%20Of%20RN6G%20In%20Subjects%20With%20Geographic%20Atrophy%20Secondary%20to%20Age-related%20Macular%20Degeneration

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04382923 2.5 mg/kg: PF-04382923 (RN6G) at 2.5 milligrams per kilogram (mg/kg) was administered as an intravenous (IV) infusion over 30 minutes every 28 days for 11 doses.
- PF-04382923 7.5 mg/kg: PF-04382923 at 7.5 mg/kg was administered as an IV infusion over 30 minutes every 28 days for 11 doses.
- PF-04382923 15.0 mg/kg: PF-04382923 at 15.0 mg/kg was administered as an IV infusion over 30 minutes every 28 days for 11 doses.
- Placebo: Placebo was administered as an IV infusion over at least 30 minutes every 28 days for 11 doses.
Period: Overall Study
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Started | 2 | 3 | 3 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 3 | 2
Not completed — Discontinued | 2 | 1 | 2 | 2
Not completed — Ongoing at Date of Cut-Off | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.5 (0.7) | 71.0 (6.2) | 74.0 (12.2) | 73.0 (11.3) | 74.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 0 | 7
  Male | 1 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction (in Study Eye) in Rate of Growth of Geographic Atrophy (GA) at Day 309
Description: GA is the advanced form of dry age-related macular degeneration (AMD). The reduction in GA area of the study eye was based on Fundus Autofluorescence (FAF) at 30 days post last dose administration (Day 309).
Time Frame: Baseline and Day 309
Population: Analysis was not performed due to early study termination. As only 10 participants enrolled at the time of termination, there were not enough subjects or data to perform meaningful analyses (8 were assigned to active drug [1 was not dosed and there was notable variability on how many doses were received by the other 7]; 2 were assigned to placebo).
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Mean Reduction (in Study Eye) in Rate of Growth of GA at Day 449 (End of Study)
Description: GA is the advanced form of dry AMD. The reduction in GA area in the study eye was based on FAF at end of study (Day 449).
Time Frame: Baseline and Day 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Best Corrected Visual Acuity (BCVA) at 9, 12, 15 Months and End of Study
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity).
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage Change From Baseline in BCVA Correct Number of Letters at 9, 12, 15 Months and End of Study
Description: as for outcome 3
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage Change From Baseline in BCVA Correct Number of Lines at Months 9, 12, 15 Months and End of Study
Description: BCVA is measured using an eye chart and is reported as the number of lines read correctly in the study eye. The lower the number of lines read correctly on the eye chart, the worse the vision (or visual acuity).
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Low Luminance Best Corrected Visual Acuity (LL-BCVA) at 9, 12, 15 Months and End of Study
Description: LL-BCVA is the measure of visual acuity under low light conditions.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage Change From Baseline in LL-BCVA Correct Number of Letters at 9, 12, 15 Months and End of Study
Description: LL-BCVA is the measure of visual acuity under low light conditions.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage Change From Baseline in LL-BCVA Correct Number of Lines at 9, 12, 15 Months and End of Study
Description: LL-BCVA is the measure of visual acuity under low light conditions.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Contrast Sensitivity at 9, 12, 15 Months and End of Study
Description: Contrast sensitivity was measured using the Pelli-Robson chart at 1 meter. Participants were tested for contrast sensitivity using +0.50 addition over the protocol refraction providing the best-corrected distance VA. Contrast sensitivity was recorded as the log of the faintest triplet for which 2 of the 3 letters were read correctly.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage Change From Baseline in Contrast Sensitivity at 9, 12, 15 Months and End of Study
Description: Contrast sensitivity was measured using the Pelli-Robson chart at 1 meter. Subjects were tested for contrast sensitivity using +0.50 addition over the protocol refraction providing the best-corrected distance VA. Contrast sensitivity was recorded as the log of the faintest triplet for which 2 of the 3 letters were read correctly.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Reading Speed at 9, 12, 15 Months and End of Study
Description: Reading speed in the study eye was assessed using modified Bailey-Lovie word charts. Participants read the chart for 2 minutes and the number of words read correctly per minute was totaled. An increase in the number of words read correctly indicated an improvement and a decrease in the number of words read correctly indicated a worsening.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Placebo in Reading Speed at 9, 12, 15 Months and End of Study
Description: as for outcome 11
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Percentage Change From Baseline in Reading Speed at 9, 12, 15 Months and End of Study
Description: as for outcome 11
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Reading Acuity at 9, 12, 15 Months and End of Study
Description: Reading Acuity was measured using the Radner reading charts and expressed in terms of logRAD (logrithmic Reading Acuity Determination).
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Placebo in Reading Acuity at 9, 12, 15 Months and End of Study
Description: Reading Acuity was measured using the Radner reading charts and expressed in terms of logRAD.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Percentage Change From Baseline in Reading Acuity at 9, 12, 15 Months and End of Study
Description: Reading Acuity was measured using the Radner reading charts and expressed in terms of logRAD.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Critical Print Size Reading at 9, 12, 15 Months and End of Study
Description: The critical print size is the smallest print size at which participants can read with their maximum reading speed.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Placebo in Critical Print Size Reading at 9, 12, 15 Months and End of Study
Description: The critical print size is the smallest print size at which participants can read with their maximum reading speed.
Time Frame: Baseline, Month 9, Month 12, Month 15, and End of Study
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Laboratory assessments include: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein); coagulation assessments.
Time Frame: Day 85 and Day 169
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Abnormal Change From Baseline in Vital Signs
Description: Vital sign assessments include: supine systolic and diastolic blood pressure, pulse rate and body temperature.
Time Frame: Screening, Days 28, 57, 85, 113, 141, and 169
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Electrocardiogram (ECG) Findings
Description: Clinically significant ECG findings include: corrected QT (QTc) > 450 msec, QTc >500 msec, change in QTc between 30 and 60 msec, change in QTc greater than or equal to 60 msec.
Time Frame: Days 28, 57, 85, 113 and 169
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA)
Description: The number of participants with positive ADA was to be summarized for each treatment arm.
Time Frame: Day 57 and Day 169
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) According to Seriousness
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Seriousness of an AE was assessed under the criteria of serious adverse event (SAE). An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Days 28, 57, 85, 113, 141 and 169
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 2 | 3 | 3 | 2
Participants
  AE | 2 | 0 | 1 | 1
  SAE | 1 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Treatment-Related TEAEs
Description: An AE was an untoward medical occurrence in a participant who received study drug without regard to causal relationship. An investigator's relationship assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an AE.
Time Frame: Days 28, 57, 85, 113, 141 and 169
Population: The safety analysis set included all participants who received at least one dose of study product.
Measure: Number; unit: Participants
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 2 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0

25. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Days 1, 28,57, 85, 169, 253, 281, 309, 337, and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Time Frame: Days 1, 28,57, 85, 169, 253, 281, 309, 337, and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero Until Last Sampling Time (AUCt)
Time Frame: Days 1, 28,57, 85, 169, 253, 281, 309, 337, and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Clearance at Steady State (CLss)
Description: Steady state total body clearance equals infusion rate (zero order) divided by steady state plasma concentration of study drug (R0/Css)
Time Frame: Days 1, 28,57, 85, 169, 253, 281, 309, 337, and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Accumulation Ratio (Rac) for AUCt
Time Frame: Days 1, 28,57, 85, 169, 253, 281, 309, 337, and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Plasma Population PK Parameters
Description: Population PK parameters were to be evaluated for Cmax, AUCt, Cmin, CLss, and Rac for AUCt between the first and last (11th) doses.
Time Frame: Days 1, 28, 57, 85, 169, 253, 281, 309, 337 and 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Change From Baseline in Total Amyloid Beta (A-Beta) 1-x Plasma Concentration at End of Study (Day 449)
Description: Concentration of total amino acid peptide, known as A-Beta 1-x, in plasma.
Time Frame: Baseline, Day 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

32. Secondary Outcome: Change From Baseline in Amyloid Beta (A-Beta) 1-40 Plasma Concentration at End of Study (Day 449)
Description: Concentration of amino acid peptide, known as A-Beta 1-40, in plasma.
Time Frame: Baseline, Day 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

33. Secondary Outcome: Change From Baseline in Amyloid Beta (A-Beta) 1-42 Plasma Concentration at End of Study (Day 449)
Description: Concentration of amino acid peptide, known as A-Beta 1-42, in plasma.
Time Frame: Baseline, Day 449
Population: as for outcome 1
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-04382923 2.5 mg/kg | PF-04382923 7.5 mg/kg | PF-04382923 15.0 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/3 | 1/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04382923 2.5 mg/kg (N=2) | PF-04382923 7.5 mg/kg (N=3) | PF-04382923 15.0 mg/kg (N=3) | Placebo (N=2)
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04382923 2.5 mg/kg (N=2) | PF-04382923 7.5 mg/kg (N=3) | PF-04382923 15.0 mg/kg (N=3) | Placebo (N=2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to an organizational decision, which was not based on safety or efficacy concerns. As only 10 participants enrolled at the time of termination, there were not enough subjects or data to perform meaningful analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.